CLINICAL TRIAL: NCT02114099
Title: An Open Label, Non-comparative Phase II Trial to Evaluate the Effects of Atorvastatin on the Persistent Coronary Arterial Aneurysm in Children With Kawasaki Disease: Safety and Efficacy
Brief Title: Trial of Atorvastatin on the Persistent Coronary Aneurysm in Children With Kawasaki Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200612128M
Record Dates: First submitted 2010-06-28; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Kawasaki Disease; Aneurysm, Coronary
Keywords: Kawasaki Disease; Aneurysm, Coronary
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Coronary Aneurysm | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atorvastatin (Experimental): prescribe Atorvastatin to see its effect
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 10 mg qd x1 year
  Other Names: Lipitor

SUMMARY:
Background Kawasaki disease (KD) is characterized by fever, bilateral nonexudative conjunctivitis, erythema of the lips and oral mucosa, changes in the extremities, rash, and cervical lymphadenopathy. Incidence of late coronary artery aneurysms or ectasia, which may lead to myocardial infarction (MI), sudden death, or ischemic heart disease, decreased after the introduction of intravenous immunoglobulin therapy. However, significant persistent coronary arterial lesions or aneurysms may still occur in about 1-3 % of the patients.

Atorvastatin (Lipitor®), a kind of statin, is a selective competitive inhibitor of 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase. This drug had been safely and widely used for treatment of adult hyperlipidemia, prevention of coronary heart disease and familial hypercholesterolemia in childhood. In addition to the cholesterol-lowering effects, statins exerts diverse cellular, cholesterol-independent effects, including improvement in endothelial function, inhibition of neurohormonal activation, and reduction in levels of proinflammatory cytokines. Based on the above concepts, some patients with infrarenal abdominal aortic aneurysms received statin therapies and then the growth rate of aneurysms slowed down.

Therefore, the investigators may hypothesize that Atorvastatin is helpful in the regression of persistent coronary lesions in KD patients due to its effect of anti-inflammation. In NTUH, there are about 20 KD patients with coronary lesions persistent for many years. And the investigators plan to conduct the clinical trial with atorvastatin to evaluate the effects of Atorvastatin on the persistent coronary arterial lesions/aneurysms in children with Kawasaki disease including safety and efficacy.

Methods

There are around 20 KD patients eligible for this study. After they sign the IRB-approved ICF, they will be enrolled for this study. Briefly, this study is divided into three stages: screening & enrollment stage (I), treatment & follow-up stage (II) for 1 year and final data analysis stage (III). Measurements include basic vital sign, electrocardiography, liver function, muscle enzyme, inflammatory markers and echocardiography.

Predicted results

1.Oral atorvastatin therapy can effectively prevent the progression of coronary lesions in KD patients.

DETAILED DESCRIPTION:
Background Kawasaki disease (KD) is characterized by fever, bilateral nonexudative conjunctivitis, erythema of the lips and oral mucosa, changes in the extremities, rash, and cervical lymphadenopathy. Incidence of late coronary artery aneurysms or ectasia, which may lead to myocardial infarction (MI), sudden death, or ischemic heart disease, decreased after the introduction of intravenous immunoglobulin therapy. However, significant persistent coronary arterial lesions or aneurysms may still occur in about 1-3 % of the patients.

Aspirin and warfarin, the recommended medication to prevent and decrease the incidence of coronary artery events, can't guarantee the coronary patency in these KD patients. Thus, it's urgent to look for an effective and safe treatment to make sure the coronary lesions will stabilize even regress gradually.

Several groups studied the clinical characteristics of KD patients with coronary sequelae and showed there was association between elevated inflammatory markers and the persistence of coronary lesions. Atorvastatin (Lipitor®), a kind of statin, is a selective competitive inhibitor of 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase. This drug had been safely and widely used for treatment of adult hyperlipidemia, prevention of coronary heart disease and familial hypercholesterolemia in childhood. In addition to the cholesterol-lowering effects, statins exerts diverse cellular, cholesterol-independent effects, including improvement in endothelial function, inhibition of neurohormonal activation, and reduction in levels of proinflammatory cytokines. Based on the above concepts, some patients with infrarenal abdominal aortic aneurysms received statin therapies and then the growth rate of aneurysms slowed down.

Therefore, the investigators may hypothesize that Atorvastatin is helpful in the regression of persistent coronary lesions in KD patients due to its effect of anti-inflammation. In NTUH, there are about 20 KD patients with coronary lesions persistent for many years. And the investigators plan to conduct the clinical trial with atorvastatin to evaluate the effects of Atorvastatin on the persistent coronary arterial lesions/aneurysms in children with Kawasaki disease including safety and efficacy.

Methods

There are around 20 KD patients eligible for this study. After they sign the IRB-approved ICF, they will be enrolled for this study. Briefly, this study is divided into three stages: screening & enrollment stage (I), treatment & follow-up stage (II) for 1 year and final data analysis stage (III). Measurements include basic vital sign, electrocardiography, liver function, muscle enzyme, inflammatory markers and echocardiography.

Predicted results

1.Oral atorvastatin therapy can effectively prevent the progression of coronary lesions in KD patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Kawasaki Disease with giant aneurysm
* Must be older than 10 years old

Exclusion Criteria:

* Subjects ever received coronary artery bypass graft (CABG) surgery.
* Subjects have active hepatitis or persistent abnormal liver function such as elevated GOT and GPT.
* Subjects have the past history of rhabdomyolysis.
* Female subjects are pregnant or plan for child-bearing during study periods.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
size of coronary aneurysm | 2 years

SECONDARY OUTCOMES:
muscle enzyme and liver function | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Tai Lin, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan